CLINICAL TRIAL: NCT01667237
Title: Feasibility of a Short Home-based Rehabilitation Program for Cancer Patients Waiting for Lung Resection Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Didier Saey, Adjunct professor, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20525
Record Dates: First submitted 2010-07-01; First posted 2012-08-17 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: Pulmonary rehabilitation program; Lung cancer; Lung resection surgery; Home-based
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pulmonary rehabilitation (Experimental)
  Interventions: Behavioral: Home-based pulmonary rehabilitation program

INTERVENTIONS:
Behavioral: Home-based pulmonary rehabilitation program — The rehabilitation program will be a self-monitored and minimally supervised home-exercise program. Exercise training modalities and intensity will be adapted to patient's individual condition. It will include aerobic and strength exercises 5 times a week for 4 weeks. Aerobic training will be done on a portable ergocycle. The target intensity will correspond to 60% of the maximal work rate achieved during the maximal progressive cardio-pulmonary exercise test, aiming for a cumulative time of 40 minutes per day. The heart rate, corresponding to an exercise level of 60% of max exercise capacity during the maximum exercise test, will be noted and patients will be instructed to train at this heart rate ± 10 beats. Muscle exercises will be performed using elastic bands and use of gravity.

SUMMARY:
The general objectives of this study are to verify the feasibility of a short home-based rehabilitation program for cancer patients prior to lung resection surgery, and to quantify its effects on aerobic capacity, exercise tolerance and skeletal muscle strength.

Therefore, the hypotheses of this study are that:

1. Implementation of a short home-based rehabilitation program (4 weeks) based on exercise training is feasible and safe in patients with lung cancer resection candidates.
2. Compared to control patients, patients included in the home-based rehabilitation program will improve significantly their aerobic capacity, exercise tolerance and arms and legs muscle force.

DETAILED DESCRIPTION:
Being the leading cause of death from cancer, lung cancer represents a pressing health issue which generates significant social costs. In Canada, in 2009, an estimated 23 400 people will be diagnosed with lung cancer, and 20 500 will die from the disease. For people with localized non small cell lung cancer (NSCLC), lung resection surgery offers the best chance of curing the disease. In addition with lung cancer, these patients often experience such effects as a reduction in their exercise capacity and tolerance, muscle weakness, and decreased quality of life. Many researches demonstrated a link between a low exercise capacity and cardiopulmonary complications surrounding surgery. Therefore, the implementation of a preoperative pulmonary rehabilitation program, focused on improving aerobic capacity, could have significant positive outcomes, notably by reducing operative risks. The effectiveness of pulmonary rehabilitation, whether carried-out in a supervised setting or as a home-based program, is well recognized and such programs are included in guidelines for many pulmonary diseases. Despite these facts, few researches have studied its impact on lung cancer patients waiting for surgery. Moreover, not one have examined the feasibility and effectiveness of a home-based program for this population.

We plan to use that time waiting for surgery to increase exercise capacity and work tolerance of cancer patients waiting for surgery. Our expertise in pulmonary rehabilitation will prove to be invaluable to carry out this research project which objectives are to verify the feasibility of a short home-based rehabilitation program for cancer patients waiting for lung resection surgery, and to measure its effects on aerobic capacity, work tolerance and muscle strength.

In this way, we hope to contribute in developing innovative interventions that will assist the Canadian Lung Association's mission of improving the health of patients with respiratory problems. The results of this study will lead toward the development of a multicenter, randomized study that will be designed to verify the impact of such interventions on postoperative complications in this population.

Experimental design:

This pilot study will take place at the research center of the Institut de cardiologie et de pneumologie de Québec (IUCPQ), in collaboration with the thoracic surgery division and the Pavillon de Prevention des Maladies Cardiaques (PPMC). Once the lung cancer and surgical procedure considered by pneumologist, we will obtain the patient's consent and we will proceed to the initial assessment.

After the initial evaluation participants will undergo a 4-week home-based rehabilitation program under the supervision of an exercise specialist certified by the American College of Sport Medicine. Patients will be reevaluated after 4 weeks.

Preliminary screening: An initial screening, including maximal oxygen consumption assessment, will be performed under the supervision of a respiratory physician (Dr F. Maltais) to ensure that patients meet the all the inclusion and exclusion criteria of the study. In addition, a brief history of each patient's disease course and medication will be recorded.

Anthropometric measurements: Weight and height will be measured to determine the Body Mass Index (BMI). Body composition will be analyzed by bio-impedance (InBody 520, Biospace).

Quality of life and psychological distress: Generic quality-of-life questionnaires provide information on many aspects of a patient's life and can also be used to discriminate between patients within the same population. However, they are not as responsive to change as disease-specific questionnaires. Thus, generic quality-of-life assessment will be obtained at the time of enrolment. The SF-36 survey was selected for its ease of administration and because it is the most largely used questionnaire. A French version of the SF-36 is currently available. These data will be obtained only for descriptive analyses.

Pulmonary function tests: Standard pulmonary function tests including spirometry, lung volumes, and carbon monoxide diffusion capacity will be obtained for all subjects during the initial evaluation, according to previously described guidelines, and related to appropriate reference values.

Incremental cycle exercise test: In order to determine peak aerobic capacity and eligibility, and to quantify changes in exercise tolerance occurring with exercise training, an incremental exercise test will be performed (before inclusion). Patients will be seated on an electrically braked ergocycle (Quinton Corival 400; A-H Robins, Seattle, WA) and connected to the exercise circuit through a mouthpiece (Sensor Medics, Vpeak Legacy, Yorba Linda, CA). A progressive stepwise exercise test will be performed up to individual's peakimum capacity, using exercise steps of 1 minute and increments of 5-10 watts. Heart rate and oxygen saturation will be recorded using pulse oximetry and ECG, respectively. Symptoms of dyspnea and leg fatigue will be recorded using a modified Borg scale for perceived exertion52. Testing will take place under medical supervision, in the exercise physiology laboratory of IUCPQ research center.

Constant workrate cycle exercise test and 6-min walking test: A constant workrate cycle exercise test and a 6-min walking test will be performed to quantify changes in exercise tolerance occurring with exercise training.

1. During the constant workrate cycle exercise test, patients will be asked to pedal at 80% max exercise work rate determined during the maximal test, and the time to exhaustion will be measured. Heart rate, dyspnea Borg score, and oxygen saturation will be monitored. Supplemental oxygen will be used if oxygen saturation < 90%.
2. For the 6-min walking test, patients will also be asked to walk as far as possible for 6 minutes with standardized encouragement53. Two trials will be done and only the best one will be used for data analysis. Monitoring of respiratory and cardiac parameters, in addition to dyspnea and leg fatigue (modified Borg scale) will be done during the test.

Strength evaluation:

1. Quadriceps strength will be assessed in two ways. First, by maximum voluntary contraction, and second, by measuring supramaximal twitch tension from a series of twitch following a magnetic stimulation (Magstim 200; Magstim Co.) of the femoral nerve as previously described. Generated force will be measured by an isometric force gauge while subjects will be in a standardized positioning. Validity and sensitivity of this equipment have previously been studied and we have used it in previous studies.
2. Maximum voluntary contraction of the biceps brachii, deltoid and hamstring will be measured with a hand-held dynamometer (Microfet. Hoggan Inc, USA), using the method described and validated by Andrews and colleagues56. Finally, a maximum prehension strength will be assessed with a hydraulic dynamometer (Jamar).

ELIGIBILITY:
Inclusion Criteria:

* Suffering from a non-small cell lung cancer on a waiting list for lung resection
* Having a VO2 Peak value of less than 20mL/kg/min.

Exclusion Criteria:

* SaO2 less less than 80% during the cardiopulmonary exercise test
* Contraindications to exercise testing (per American Thoracic Society/American College of Chest Physicians Exercise Testing Guidelines)
* A history of significant or cardiovascular disease, hypertension, diabetes, or musculoskeletal concerns that might limit the ability of these subjects to perform active exercises
* Severe psychiatric illness compromising training rehabilitation observance

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
To verify the feasability of a short home-based rehabilitation for cancer patients prior to lung resection surgery program. | During a 4 week rehabilitation programs preceeding surgery

SECONDARY OUTCOMES:
To quantify the cycle endurance change induced by a short home-based rehabilitation for cancer patients prior to lung resection surgery program. | before and after a 4 week rehabilitation programs preceeding surgery
To quantify the quadriceps muscle force change induced by a short home-based rehabilitation for cancer patients prior to lung resection surgery program. | before and after a 4 week rehabilitation programs preceeding surgery

CONTACTS AND LOCATIONS:
Overall Officials: Didier Saey, Phd., Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- CRIUCPQ, Québec, Quebec, Canada